CLINICAL TRIAL: NCT03801694
Title: To Evaluate the Role of Plasma Catecholamine Levels in Predicting the Development of Myocardial Depression in Acute Neurological Patients
Brief Title: Predicting the Development of Myocardial Depression in Acute Neurological Patients
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Tamara Strohm, Assistant Professor- Neurology, Ohio State University
Other Study IDs: 2018H0436
Record Dates: First submitted 2019-01-03; First posted 2019-01-11 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Myocardial Depression; Takotsubo Syndrome; Subarachnoid Hemorrhage; Acute Ischemic Stroke
MeSH Terms: conditions — Takotsubo Cardiomyopathy; Subarachnoid Hemorrhage; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Baseline plasma catecholamine levels, transthoracic ECHO(TTE), Troponin T, EKG and BNP will be obtained. Thereafter, we will follow daily plasma catecholamine levels, troponin, EKG and BNP up to 5 days from the study onset
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess the levels of serum catecholamines associated with myocardial depression (MD) in patients with acute neurological injury.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the level of plasma catecholamines, associated with myocardial depression (MD) as noted on Transthoracic ECHO (TTE) by evidence of wall motion abnormalities (WMA) with or without drop in ejection fraction or symptomatic heart failure (HF). Takotsubo syndrome (TTS) is commonly diagnosed after the onset of HF once patients become symptomatic. The investigators intend to study whether early MD can be detected by identifying certain levels of plasma catecholamines and whether the level correlates with severity of myocardial depression. Identification of early MD changes can lead to alteration of management strategies and may help prevent worsening of HF. Highly selected patients with Subarachnoid Hemorrhage (SAH) or Acute Ischemic Stroke (AIS) requiring induced hypertension with the use of norepinephrine infusion will be recruited to enroll in this pilot study. This group of patients are expected to have high circulating catecholamines and are more likely to develop MD. Given the prevalence of TTS in females and elderly, 10 female patients >50 years admitted to the neuro ICU with diagnosis of either AIS or SAH will be enrolled. Patients with history of coronary artery disease, smoking, poorly controlled diabetes with HbA1c >8 and uncontrolled hypertension will be excluded. Patients with poor ECHO windows will also be excluded. Baseline plasma catecholamine levels, transthoracic ECHO(TTE), Troponin T, EKG and BNP will be obtained and will be followed daily through the study duration.

ELIGIBILITY:
Inclusion Criteria:

* female patients >50 years admitted to the neuro ICU with diagnosis of either acute ischemic stroke or subarachnoid hemorrhage
* Only patients predicted to be on norepinephrine infusion for at least 48 hrs will be selected.

Exclusion Criteria:

* patients with known history of heart failure will be excluded
* Patients with history of coronary artery disease, smoking, poorly controlled diabetes with HbA1c >8 and uncontrolled hypertension will be excluded.
* Patients with poor ECHO windows will be excluded

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female patients >50 years admitted to the neuro ICU with diagnosis of either acute ischemic stroke or subarachnoid hemorrhage
Study Population: Highly selected partients with Subarachnoid Hemorrhage (SAH) or Acute Ischemic Stroke (AIS) requiring induced hypertension with the use of norepinephrine infusion will be involve in this pilot study.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2024-04-14 (Actual); Study Completion 2024-04-14 (Actual)

PRIMARY OUTCOMES:
Association of plasma catecholamine levels with stress induced cardiomyopathy | up to 5 days
  Baseline plasma catecholamine levels as well as daily levels will be measured until up to 5 days from study onset. Baseline transthoracic ECHO followed by daily ECHO with strain imaging will be obtained to assess for evidence of myocardial depression. The investigators will assess the correlation of plasma catecholamine levels (i.e level of dopamine, epinephrine and norepinephrine) in the development of myocardial depression. In other words, the investigators will evaluate the level of catecholamines that is associated with stress induced cardiomyopathy. If participants develop symptomatic heart failure before 5 days, study will stop at that point.
Association of troponin levels with stress induced cardiomyopathy | up to 5 days
  Baseline troponin level will be measured as well as daily levels will be obtained for 5 days. The investigators will study the correlation of troponin levels with the myocardial depression noted on ECHO.

SECONDARY OUTCOMES:
Association of ST-T changes on EKG with stress induced cardiomyopathy | up to 5 days
  Baseline EKG and daily EKG measurements will be taken. These will be examined for ST-T wave changes in participants with evidence of myocardial depression on ECHO.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Strohm, Principal Investigator — Ohio State University
Locations (1):
- The Ohio Sate University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No